CLINICAL TRIAL: NCT00101114
Title: A Phase II Study of the RAF-Kinase Inhibitor BAY 43-9006 (NSC-724772, IND-69,896) in Combination With Interferon-Alpha 2B in Patients With Advanced Renal Cancer
Brief Title: Sorafenib and Interferon Alfa in Treating Patients With Metastatic or Unresectable Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-03061; S0412; U10CA032102 (NIH); CDR0000405893 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2005-01-07; First posted 2005-01-10 (Estimated); Last update posted 2013-02-28 (Estimated); Status verified 2013-02

CONDITIONS: Clear Cell Renal Cell Carcinoma; Recurrent Renal Cell Cancer; Stage III Renal Cell Cancer; Stage IV Renal Cell Cancer
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib; Introns

ARMS (1):
- Treatment (sorafenib tosylate, interferon alpha-2b) (Experimental): Patients receive oral sorafenib twice daily on days 1-28 and interferon alfa subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: sorafenib tosylate; Biological: recombinant interferon alfa-2b; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: sorafenib tosylate — Given PO
  Other Names: BAY 43-9006; BAY 43-9006 Tosylate Salt; BAY 54-9085; Nexavar; SFN
Biological: recombinant interferon alfa-2b — Given SC
  Other Names: Alfatronol; Glucoferon; Heberon Alfa; IFN alpha-2B; Intron A
Other: laboratory biomarker analysis — Optional correlative studies

SUMMARY:
This phase II trial is studying how well giving sorafenib with interferon alfa works in treating patients with metastatic or unresectable kidney cancer. Sorafenib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Interferon alfa may interfere with the growth of tumor cells and slow the growth of kidney cancer. Sorafenib may help interferon alfa work better by making tumor cells more sensitive to the drug

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess response (confirmed complete and partial responses) of patients with advanced renal cell cancer treated with the combination of BAY-43-9006 and interferon alfa-2b.

SECONDARY OBJECTIVES:

I. To assess the probability of treatment failure at 6 months and the median overall survival of this group of patients.

II. To evaluate the quantitative and qualitative toxicities of this regimen. III. To investigate in a preliminary manner the association of tumor response with measures of increased signaling through the Ras-Raf pathway (p-MAPK, p-JNK, p-p38, and p-AKT), with VHL gene status, and whether changes in levels of IL-6 and tumor markers of hypoxia including PAI-1, VEGF, and osteopontin correspond with clinical outcomes.

OUTLINE: This is a multicenter study.

Patients receive oral sorafenib twice daily on days 1-28 and interferon alfa subcutaneously on days 1, 3, 5, 8, 10, 12, 15, 17, 19, 22, 24, and 26. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for 1 year and then every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed renal cell carcinoma which is either metastatic (M1) or unresectable (M0); patients must have a component of conventional clear cell renal carcinoma; patients with true papillary renal cell carcinoma, sarcomatoid features without any clear cell component, chromophobe, oncocytoma, collecting duct tumors and transitional cell carcinoma are NOT eligible
* Patients must have measurable disease; soft tissue disease, which has been radiated in the 2 months prior to registration, is not assessable as measurable disease; X-rays, scans, or physical examinations used for tumor measurement must have been completed within 28 days prior to registration; X-rays, scans or physical examinations for non-measureable disease must have been completed within 42 days prior to registration; all disease must be assessed
* Patients with metastatic disease who have a resectable primary tumor and are deemed a surgical candidate may have undergone resection and have recovered from surgery; at least 28 days must have elapsed since surgery and patient must have recovered from any adverse effects of surgery
* Patients must not have received any prior systemic therapy for renal cell carcinoma, including chemotherapy, interferon, interleukin-2, other biologic response modifiers, anti-angiogenic therapy, hormonal therapy, or any other experimental systemic therapy; prior treatment with thyroid medications is allowed
* Patients may have received prior radiation therapy to less than 25% of the bone marrow; at least 28 days must have elapsed since completion of prior radiation therapy; patients must have recovered from all associated toxicities at the time of registration
* Total bilirubin =< institutional upper limit of normal
* SGOT or SGPT =< 2.5 x institutional upper limit of normal
* Serum creatinine =< institutional upper limit of normal or calculated creatinine clearance >= 60 mL/min for patients with creatinine levels above institutional normal

  * Patients who have had a prior nephrectomy must have a serum creatinine =< 2 x institutional upper limit of normal
* Patients must be offered the opportunity to consent for specimen submission
* Patients must have a Zubrod performance status of 0-1
* Patients with a history of brain metastases or who currently have treated to untreated brain metastases are not eligible; patients with clinical suspicion of brain metastases must have a brain CT or MRI negative for metastatic disease obtained within 56 days prior to registration and must not have any new symptoms since radiographic evaluation was done
* Any ongoing requirement for systemic corticosteroid therapy is not permitted; topical and/or inhaled steroids are allowed
* Patients must not be on drugs known to be potent inhibitors of the CYP 3A4 enzyme as BAY 43-9006 is at least partially metabolized by this enzyme in the liver; the possible effect that inhibitors of this enzyme may have on the metabolism of BAY 43-9006 is unknown; therefore, patients who are on the following drugs are not eligible (patients should not take these drugs while receiving protocol treatment): ketoconazole, itraconazole, ritonavir, products containing grapefruit juice, cyclosporine, carbamazepine, phenytoin and phenobarbital)
* Patients must be able to take oral medication without crushing, dissolving or chewing tablets
* The effects of BAY 43-9006 on the developing human fetus at the recommended therapeutic dose are unknown; for this reason and because raf kinase inhibitor agents as well as other therapeutic agents used in this trial are known to be teratogenic, patients must not be pregnant or nursing; women/men of reproductive potential must have agreed to use an effective contraceptive method (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* No other prior malignancy is allowed except for the following: adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, adequately treated Stage I or II cancer from which the patient is currently in complete remission, or any other cancer from which the patient has been disease-free for 5 years
* If Day 28, 42, or 56 falls on a weekend or holiday, the limit may be extended to the next working day
* All patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines
* At the time of patient registration, the treating institution's name and ID number must be provided to the Data Operations Center in Seattle in order to ensure that the current (within 365 days) date of institutional review board approval for this study has been entered into the database

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2004-09; Primary Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Response probability | Up to 3 years

SECONDARY OUTCOMES:
Time to treatment failure | From date of registration to date of first observation of progressive disease, death due to any cause, symptomatic deterioration, or early discontinuation of treatment, assessed up to 3 years
Survival | Up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Ryan, Principal Investigator — SWOG Cancer Research Network
Locations (1):
- Southwest Oncology Group, San Antonio, Texas, United States